CLINICAL TRIAL: NCT05705297
Title: Intracardiac Echocardiography Guided Slow Pathway Cryoablation for Treatment of Atrio-ventricular Nodal Reentry Tachycardia
Brief Title: Intracardiac Echocardiography Guided Slow Pathway Cryoablation
Status: Enrolling by invitation | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, MD, University Medical Centre Ljubljana
Other Study IDs: ICE cryo AVNRT
Record Dates: First submitted 2023-01-16; First posted 2023-01-30 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Atrioventricular Nodal Reentry Tachycardia
Keywords: atrioventricular nodal reentry tachycardia; cryoablation; intracardiac echocardiography
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrioventricular nodal reentry tachycardia is best treated with catheter ablation aimed at disruption of conduction of the slow pathway. There are currently two possible options for this ablation: radiofrequency ablation and cryoablation. The first seems to result in superior success rate, however carries a small risk of collateral damage of the heart conduction system, specifically the atrioventricular (AV) node. Cryoablation seems less effective, but safer as AV nodal damage can be avoided. The aim of this study is to prospectively test possible improved efficcacy of cryoablation of the slow pathway with the use intraprocedural intracardiac echocardiography.

DETAILED DESCRIPTION:
We will prospectively enroll all patients that will be referred to our center for ablation of supraventricular tachycardia and will have an electrophysiologically proven atrioventricular nodal reentry tachycardia. In order to prove the mechanism specific maneuvers will be performed during induced sustained tachycardia. Navigation in the heart will be performed in a fluoroless fashion, with the use of a three-dimensional electro-anatomic mapping (3DEAM) system. Detailed anatomical definition and navigation in the area of the Koch triangle will be done with intracardiac echocardiography (ICE). Also, in sinus rhythm, when present, the Jackman potential will be tagged on the 3DEAM map. Cryomapping will be performed at the presumed location of the slow pathway (position of the Jackman potential or only anatomical location as defined with ICE) during ongoing tachycardia with the aim to terminate it and continue with cryoablation at the successful site.

Noninducibility will be tested with programmed and fast atrial stimulation. Patients will be followed clinically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* ECG or holter ECG evidence of regular narrow QRS complex tachycardia, intraprocedural pacing maneuvers in sinus rhythm and during ongoing tachycardia indicating presence of AVNRT

Exclusion Criteria:

* terminal or severe medical condition with expected survival of less then 12 months, deep venous thrombosis preventing access to the femoral vein, intracardiac thrombi, anatomical irregularities of pelvic veins and/or inferior vena cava, inability to induce AVNRT after the initial induction and diagnosis - enables exclusion of procedures where accidental mechanical termination of slow pathway conduction with the cryoablation catheter occurs

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult and pediatric patients with the body weight above 15 kg with documented regular narrow QRS complex tachycardia referred for catheter ablation in accordance with current guidelines (EHRA, AEPC and/or HRS).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-07-03 (Estimated)

PRIMARY OUTCOMES:
Noninducibility at the end of procedure | up to 1 day
  Noninducibility of AVNRT after cryoablation with programmed and fast atrial stimulation
Arrhythmia free survival | 12 months
  Absence of AVNRT episodes during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Matevž Jan, MD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425
- [Background] Drago F, Calvieri C, Russo MS, Remoli R, Pazzano V, Battipaglia I, Gimigliano F, Allegretti G, Silvetti MS. Low-voltage bridge strategy to guide cryoablation of typical and atypical atrioventricular nodal re-entry tachycardia in children: mid-term outcomes in a large cohort of patients. Europace. 2021 Feb 5;23(2):271-277. doi: 10.1093/europace/euaa195. PMID 33038208
- [Background] Pandozi C, Lavalle C, Bongiorni MG, Catalano A, Pelargonio G, Russo M, Piro A, Carbone A, Narducci ML, Galeazzi M, Ficili S, Piccolo F, Maddaluno F, Malacrida M, Colivicchi F, Segreti L. High-density mapping of Koch's triangle during sinus rhythm and typical AV nodal reentrant tachycardia: new insight. J Interv Card Electrophysiol. 2021 Sep;61(3):487-497. doi: 10.1007/s10840-020-00841-8. Epub 2020 Aug 6. PMID 32766944
- [Background] Brugada J, Blom N, Sarquella-Brugada G, Blomstrom-Lundqvist C, Deanfield J, Janousek J, Abrams D, Bauersfeld U, Brugada R, Drago F, de Groot N, Happonen JM, Hebe J, Yen Ho S, Marijon E, Paul T, Pfammatter JP, Rosenthal E; European Heart Rhythm Association; Association for European Paediatric and Congenital Cardiology. Pharmacological and non-pharmacological therapy for arrhythmias in the pediatric population: EHRA and AEPC-Arrhythmia Working Group joint consensus statement. Europace. 2013 Sep;15(9):1337-82. doi: 10.1093/europace/eut082. Epub 2013 Jul 12. PMID 23851511
- [Result] Santangeli P, Proietti R, Di Biase L, Bai R, Natale A. Cryoablation versus radiofrequency ablation of atrioventricular nodal reentrant tachycardia. J Interv Card Electrophysiol. 2014 Mar;39(2):111-9. doi: 10.1007/s10840-013-9842-2. Epub 2013 Nov 29. PMID 24293174
- [Result] Deisenhofer I, Zrenner B, Yin YH, Pitschner HF, Kuniss M, Grossmann G, Stiller S, Luik A, Veltmann C, Frank J, Linner J, Estner HL, Pflaumer A, Wu J, von Bary C, Ucer E, Reents T, Tzeis S, Fichtner S, Kathan S, Karch MR, Jilek C, Ammar S, Kolb C, Liu ZC, Haller B, Schmitt C, Hessling G. Cryoablation versus radiofrequency energy for the ablation of atrioventricular nodal reentrant tachycardia (the CYRANO Study): results from a large multicenter prospective randomized trial. Circulation. 2010 Nov 30;122(22):2239-45. doi: 10.1161/CIRCULATIONAHA.110.970350. Epub 2010 Nov 15. PMID 21098435
- [Result] Rodriguez-Entem FJ, Exposito V, Gonzalez-Enriquez S, Olalla-Antolin JJ. Cryoablation versus radiofrequency ablation for the treatment of atrioventricular nodal reentrant tachycardia: results of a prospective randomized study. J Interv Card Electrophysiol. 2013 Jan;36(1):41-5; discussion 45. doi: 10.1007/s10840-012-9732-z. Epub 2012 Oct 19. PMID 23080326